CLINICAL TRIAL: NCT00338377
Title: Lymphodepletion Plus Adoptive Cell Transfer With or Without Dendritic Cell Immunization in Patients With Metastatic Melanoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Prometheus Laboratories (Industry); Key Biologics, LLC (Industry); National Cancer Institute (NCI) (NIH); Adelson Medical Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0069; NCI-2012-01368 (Registry Identifier: NCI CTRP); 5R01CA187076-02 (NIH)
Record Dates: First submitted 2006-02-10; First posted 2006-06-20 (Estimated); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Melanoma
Keywords: Melanoma; Regional nodal disease; Dendritic Cell Immunization; Lymphodepletion; Adoptive Cell Transfer; T Cells; Vaccine; Cyclosphosphamide; Cytoxan; Neosar; Dendritic Cells; Tumor Infiltrating Lymphocytes; TIL Cells; MART Peptide; Fludarabine; Fludarabine Phosphate; Fludara; Proleukin; IL-2; Interleukin-2; Leptomeningeal disease
MeSH Terms: conditions — Melanoma; Meningeal Neoplasms | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate; Interleukin-2; aldesleukin; Mesna

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Group A: Chemotherapy + IL-2 plus T-cells (Experimental): Cyclophosphamide 60 mg/kg/d by vein (IV) over 2 hours Days -7 and -6 (with Mesna) and Fludarabine 25 mg/m^2 IV daily Days -5 to -1 before T cell infusion. On Day 0, up to 1.5 x 10^11 T cells IV infusion over 30-60 minutes. Interleukin-2 12-16 hours after T cell infusion at standard dose of 720,000 IU/kg as intravenous bolus over 15 minute period every 8-16 hours for up to 15 doses on Days 1-5 and 22-26.
  Group A has been closed to new patient entry as of January 14, 2016.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: T-Cells; Biological: Interleukin-2; Drug: Mesna
- Group B: Chemotherapy + IL-2 plus T-Cells + Vaccine (Experimental): Chemotherapy and IL-2 plus T-cells and the vaccine of dendritic cells received by vein (IV) about 4 hours after T-cells and again on Day 21 (+/- 7 days). Cyclophosphamide 60 mg/kg/d IV over 2 hours Days -7 and -6 (with Mesna) and Fludarabine 25 mg/m^2 IV daily Days -5 to -1 before T cell infusion. On Day 0, up to 1.5 x 10^11 T cells IV infusion over 30-60 minutes. Interleukin-2 12-16 hours after T cell infusion at standard dose of 720,000 IU/kg as intravenous bolus over 15 minute period every 8-16 hours for up to 15 doses on Days 1-5 and 22-26.
  Interventions: Biological: Dendritic Cell Immunization; Drug: Cyclophosphamide; Drug: Fludarabine; Biological: T-Cells; Biological: Interleukin-2; Drug: Mesna
- Group C: Prior Treatment with BRAF Inhibitor (Experimental): Chemotherapy and IL-2 plus T-cells and the vaccine of dendritic cells received by vein (IV) about 4 hours after T-cells and again on Day 21 (+/- 7 days). Cyclophosphamide 60 mg/kg/d IV over 2 hours Days -7 and -6 (with Mesna) and Fludarabine 25 mg/m^2 IV daily Days -5 to -1 before T cell infusion. On Day 0, up to 1.5 x 10^11 T cells IV infusion over 30-60 minutes. Interleukin-2 12-16 hours after T cell infusion at standard dose of 720,000 IU/kg as intravenous bolus over 15 minute period every 8-16 hours for up to 15 doses on Days 1-5 and 22-26.
  Interventions: Biological: Dendritic Cell Immunization; Drug: Cyclophosphamide; Drug: Fludarabine; Biological: T-Cells; Biological: Interleukin-2; Drug: Mesna
- Group D: Leptomeningeal Disease (Experimental): T-cells: 5.0x109 TIL administered on Day 1 and 10x109 TIL on Day 15.
  IL-2: 1.2 MIU of IL- 2 on Days 2, 4, 9, 11, 16 and 18 as tolerated. After this period, patient receives twice weekly IL-2 that will be gradually changed to weekly IL-2. After 4-6 weeks, patients switched to IL-2.
  Interventions: Biological: Intrathecal T-Cells; Biological: Intrathecal Interleukin-2
- Group E: Chemotherapy + IL-2 plus T-Cells + Vaccine (Experimental): Chemotherapy and IL-2 plus T-cells and the vaccine of dendritic cells received by vein (IV) about 4 hours after T-cells and again on Day 21 (+/- 7 days). Cyclophosphamide 60 mg/kg/d IV over 2 hours Days -7 and -6 (with Mesna) and Fludarabine 25 mg/m^2 IV daily Days -5 to -1 before T cell infusion. On Day 0, up to 1.5 x 10^11 T cells IV infusion over 30-60 minutes. Interleukin-2 12-16 hours after T cell infusion at standard dose of 720,000 IU/kg as intravenous bolus over 15 minute period every 8-16 hours for up to 15 doses on Days 1-5 and 22-26.
  Interventions: Biological: Dendritic Cell Immunization; Drug: Cyclophosphamide; Drug: Fludarabine; Biological: T-Cells; Biological: Interleukin-2; Drug: Mesna

INTERVENTIONS:
Biological: Dendritic Cell Immunization — 1x10^7 to 2.5x10^8 MART-1 peptide-pulsed Dendritic Cells given by vein over 20-30 minutes approximately 4 hrs after receiving T cells.
  Arms: Group B: Chemotherapy + IL-2 plus T-Cells + Vaccine; Group C: Prior Treatment with BRAF Inhibitor; Group E: Chemotherapy + IL-2 plus T-Cells + Vaccine
Drug: Cyclophosphamide — 60 mg/kg/d by vein over 2 hours on Days -7 and -6 before T cell infusion
  Other Names: Cytoxan; Neosar
  Arms: Group A: Chemotherapy + IL-2 plus T-cells; Group B: Chemotherapy + IL-2 plus T-Cells + Vaccine; Group C: Prior Treatment with BRAF Inhibitor; Group E: Chemotherapy + IL-2 plus T-Cells + Vaccine
Drug: Fludarabine — 25 mg/m^2 by vein daily over 30 minutes on Days -5 to -1 before T cell infusion.
  Other Names: Fludarabine Phosphate; Fludara
  Arms: Group A: Chemotherapy + IL-2 plus T-cells; Group B: Chemotherapy + IL-2 plus T-Cells + Vaccine; Group C: Prior Treatment with BRAF Inhibitor; Group E: Chemotherapy + IL-2 plus T-Cells + Vaccine
Biological: T-Cells — On Days 0, up to 1.5 x 10^11 T-cells by vein infusion over 30-60 minutes.
  Arms: Group A: Chemotherapy + IL-2 plus T-cells; Group B: Chemotherapy + IL-2 plus T-Cells + Vaccine; Group C: Prior Treatment with BRAF Inhibitor; Group E: Chemotherapy + IL-2 plus T-Cells + Vaccine
Biological: Interleukin-2 — 12-16 hours after completing the T cell infusion, all will receive high dose IL-2 on an inpatient basis at the standard dose of 720,000 IU/kg as an intravenous bolus over approximately a 15 minute period every 8-16 hours for up to 15 doses on Days 1-5 and 22-26 (+/- 7 days), as tolerated.
  Other Names: IL-2; Proleukin
  Arms: Group A: Chemotherapy + IL-2 plus T-cells; Group B: Chemotherapy + IL-2 plus T-Cells + Vaccine; Group C: Prior Treatment with BRAF Inhibitor; Group E: Chemotherapy + IL-2 plus T-Cells + Vaccine
Drug: Mesna — 60 mg/kg with D5W or NS at 125 ml/hr infused intravenously over 24 hours on Day -7 and -6.
  Other Names: Sodium 2-mercaptoethanesulfonate; Mesnum; Mesnex; NSC-113891
  Arms: Group A: Chemotherapy + IL-2 plus T-cells; Group B: Chemotherapy + IL-2 plus T-Cells + Vaccine; Group C: Prior Treatment with BRAF Inhibitor; Group E: Chemotherapy + IL-2 plus T-Cells + Vaccine
Biological: Intrathecal T-Cells — 5.0x10^9 T-cells administered on Day 1, and 10x10^9 T-cells on Day 15. 1.2 MIU of IL- 2 on Day 2, 4, 9, 11, 16 and 18 as tolerated.
  Arms: Group D: Leptomeningeal Disease
Biological: Intrathecal Interleukin-2 — 1.2 MIU of IL- 2 on Day 2, 4, 9, 11, 16 and 18 as tolerated. Then, patient receives twice weekly IL-2 that will be gradually changed to weekly IL-2. After 4-6 weeks patients switched to IL-2 maintenance.
  Other Names: IL-2
  Arms: Group D: Leptomeningeal Disease

SUMMARY:
Objectives:

The primary objective will be to determine whether patients receiving the combination of dendritic cells and high dose IL-2 (Cohort A) have sustained persistence of infused T cells compared to patients treated with T cells and high dose IL-2 alone.

Secondary endpoints will include evaluations for tumor response and studies to determine whether dendritic cells enhance the infused T cells in anti-tumor activity and their ability to migrate to the tumor site. In addition, we will evaluate the characteristics of the infused T cells that correspond with effectiveness in vivo.

Additionally, secondary objectives will include correlation of clinical parameters with survival (overall survival and progression-free survival) for all cohorts.

COHORT C

In a separate cohort (Cohort C) the primary endpoint will be the overall response rate of TIL treatment for patients who have not achieved PR or CR or have progressive disease from treatment of the BRAF inhibitor alone.

COHORT D

The primary objective of Cohort D is to confirm the safety of adoptively transferred, TIL into the CSF.

The secondary objective is the evaluation of clinical imaging and CSF response. Correlative objectives will assess if the intrathecally-infused T cells persist in the CSF, assess circulating tumor cells in the CSF, and assess various cytokine and other analyses,as feasible.

COHORT E

The primary objective of Cohort E is to determine the overall response rate of TIL treatment with cells grown by the TIL 3.0 pre-REP (Turnstile 1) phase of cellular growth.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have metastatic melanoma, uveal melanoma or stage III in-transit or regional nodal disease. (Turnstile I)
2. Patients must receive an MRI/CT of the brain or PET/CT within 6 months of consenting. If new lesions are present, PI or his designee should make final determination regarding enrollment. (Turnstile I)
3. Age greater than or equal to 12 years. (Turnstile I)
4. Clinical performance status of ECOG 0-2. (Turnstile I)
5. Patients previously treated with immunotherapy, targeted therapy, or no therapy will be eligible. Patients receiving cytotoxic agents will be evaluated by the PI or his designee as to suitable eligibility. (Turnstile I)
6. Patients must be HLA-A2 for cohort A. (Turnstile II-Chemotherapy/Cell Infusion-Inclusion Criteria)
7. Patients must have adequate TIL available. (Turnstile II)
8. Patients must have measurable metastatic melanoma. (Turnstile II - Chemotherapy/Cell Infusion -Inclusion Criteria).
9. Patients may have brain lesions which measure </= 1cm each. Lesions that are >1 cm that have been treated with SRS and in the opinion of the PI or his designee no longer represents active disease will also be allowed. (Turnstile II - Chemotherapy/Cell Infusion- Inclusion Criteria).
10. Patients of both genders must practice birth control for four months after receiving the preparative regimen. (Turnstile II - Chemotherapy/Cell Infusion- Inclusion Criteria).
11. Patients must have a documented negative pregnancy test (urine or serum) for women who have menstruation in the past 12 months and without sterilization surgery.
12. Unless surgically sterile by bilateral tubal ligation or vasectomy of partner(s), the patient agrees to continue to use a barrier method of contraception throughout the study such as: condom, diaphragm, hormonal, IUD, or sponge plus spermicide. Abstinence is an acceptable form of birth control. (Turnstile II)
13. Pregnancy testing will be performed within 7 days prior to treatment. (Turnstile II)
14. Clinical performance status of ECOG 0 - 2 at the time of chemotherapy infusion. (Turnstile II - Chemotherapy/Cell Infusion-Inclusion Criteria).
15. Absolute neutrophil count greater than or equal to 750/mm3. (Turnstile II - Chemotherapy/Cell Infusion- Inclusion Criteria).
16. Platelet count greater than or equal to 75,000/mm3. (Turnstile II - Chemotherapy/Cell Infusion- Inclusion Criteria).
17. Hemoglobin greater than or equal to 8.0 g/dl. (Turnstile II - Chemotherapy/Cell Infusion).
18. Serum ALT less than three times the upper limit of normal. (Turnstile II - Chemotherapy/Cell Infusion- Inclusion Criteria).
19. Serum creatinine less than or equal to 1.6 mg/dl. (Turnstile II - Chemotherapy/Cell Infusion-Inclusion Criteria).
20. Total bilirubin less than or equal to 2.0 mg/dl, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dl. (Turnstile II - Chemotherapy/Cell Infusion - Inclusion Criteria).
21. Patients in Cohort A will be randomized to receive either TIL alone or TIL plus Dendritic cells.
22. A stress cardiac test (stress thallium, stress MUGA, dobutamine echocardiogram or other stress test that will rule out cardiac ischemia) within 6 months of lymphodepletion. (Turnstile II - Chemotherapy/Cell Infusion-Inclusion Criteria).
23. Pulmonary function tests (FEV1>65% or FVC>65%of predicted) within 6 months of lymphodepletion. (Turnstile II - Chemotherapy/Cell Infusion - Inclusion Criteria).
24. MRI/CT of the brain within 42 days of lymphodepletion. CT scan of chest/abdomen/pelvis or PET/CT within 30 days of lymphodepletion. Exception: Patients randomized to receive dendritic cells may have an MRI of the brain within 30 days of lymphodepletion. (Turnstile II-Chemotherapy/Cell Infusion-Inclusion Criteria)
25. Patients must be receiving a B-RAF inhibitor and failed to achieve PR or CR or have progressive disease in response to B-RAF treatment (Cohort C).
26. i. Patients with MRI evidence of LMD, with or without evidence of malignant cells in CSF ("positive cytology"), or ii. Patients with evidence of malignant cells in the CSF (positive cytology), with or without MRI evidence of LMD, or iii. Patients with surgically-proven LMD (leptomeningeal involvement on pathology review) +/- MRI or CSF evidence by MRI or CSF cytology (Cohort D)
27. a. Many patients present with concomitant systemic disease outside of the central nervous system. Extra-CNS disease status should meet the following criteria: i. Patients with concomitant systemic disease under control with current or prior systemic treatment, as per primary treating physician ii. Patients without any evidence of systemic disease, either receiving systemic treatment or on active observation (Cohort D)
28. c. Previous Therapies i. Patients who are currently being treated with IT IL-2 for LMD are eligible. No wash out period is required. ii. Patients who have been previously treated with other IT therapies are eligible, as long as there is at least a 2 week wash out period iii. Patients who have previously received therapy with systemic TIL therapy are eligible.
29. (contd #28) iv. Patients with VP shunts must have VP shunts with on/off valves and must be expected to tolerate VP shunt valve off for more than 6 hours Patients who have received CNS irradiation, including whole brain radiation or stereotactic radiosurgery, are eligible, if they are at least 1 weeks post CNS-irradiation (Cohort D)Patients who are currently being treated with IT IL-2 for LMD are eligible. No wash out period is required. (Cohort D)
30. d. Other Requirements i. Patients must be able to give informed consent ii. Patients must have ECOG performance status 0, 1 or 2 and/or KPS > 50 iii. Patients must be able to swallow iv. Patients must be able to sit up with or without assistance v. Patients must be able to undergo contrast-enhanced MRI. (Cohort D)

Exclusion Criteria:

1. Has had prior systemic cancer cytotoxic chemotherapy within the past four weeks at the time of the start of the lymphodepletion regimen.
2. Has had prior B-RAF or MEK targeted therapy within 7 days prior to the start of the lymphodepletion regimen (Cohort A and Cohort B).
3. Is not receiving B-RAF treatment (Cohort C) (Turnstile II - Chemotherapy/Cell Infusion Exclusion Criteria)
4. Achieves PR or CR in response to B-RAF treatment (Cohort C).
5. Women who are pregnant or nursing will be excluded because of the potentially dangerous effects of the preparative chemotherapy on the fetus. (Turnstile II - Chemotherapy/Cell Infusion Exclusion Criteria)
6. Any active systemic infections requiring intravenous antibiotics, coagulation disorders or other major medical illnesses of the cardiovascular, respiratory or immune system, such as abnormal stress test and/or abnormal PFT. PI or his designee shall make the final determination regarding appropriateness of enrollment.(Turnstile II - Chemotherapy/Cell Infusion Exclusion Criteria)
7. Any form of primary or secondary immunodeficiency. Must have recovered immune competence after chemotherapy or radiation therapy as evidenced by lymphocyte counts (> 500/mm3), WBC (> 3,000/mm3) or absence of opportunistic infections. (Turnstile II - Chemotherapy/Cell Infusion Exclusion Criteria)
8. Require steroid therapy or steroid-containing compounds, or have used systemic steroids in the past 30 days, or have used topical or inhalational steroids in the past 2 weeks prior to lymphodepletion. Exception: Patients on physiologic dose of steroid (Turnstile II - Chemotherapy/Cell Infusion Exclusion Criteria)
9. Presence of a significant psychiatric disease, which in the opinion of the principal investigator or his designee, would prevent adequate informed consent or render immunotherapy unsafe or contraindicated. (Turnstile II - Chemotherapy/Cell Infusion Exclusion Criteria)
10. Patients with rapidly advancing systemic disease, especially those without good options of systemic treatment for their disease outside the CNS. (Cohort D)
11. Patients with rapidly advancing parenchymal brain metastases (Cohort D)
12. Pregnant patients (Cohort D)
13. Patients with rapid decline in neurological function as documented on exam and/or as per clinical judgment of treating physician (Cohort D)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1230 (Actual)
Dates: Start 2006-02-01 (Actual); Primary Completion 2030-02-28 (Estimated); Study Completion 2030-02-28 (Estimated)

PRIMARY OUTCOMES:
Objective Response (OR) | Clinical Evaluation during first 70 Days, CT Scan at 6-8 weeks (+/- 7 days) after cell infusion.
  Objective response (OR) defined as immune-related Best Overall Response (irBOR). irBOR is best confirmed immune-related response criteria (irRC) overall response over the study as a whole, recorded between the date of first dose until the last tumor assessment before subsequent therapy (except for local palliative radiotherapy for painful bone lesions) for the individual subjects in the study.
Longitudinal Immune Response in Cohort D | 4 weeks
  Longitudinal immune response defined as: Conversion of positive to negative cytology. Any perceptible improvement of the MRI findings confirmed by radiologist and/or the investigator confirmed by 2 successive MRIs 4 weeks apart. Any clinical improvement in terms of neurological symptoms.
Overall response rate (ORR) of TIL generated with the TIL 3.0 pre-REP methodology in Cohort E | At about 6 weeks and at 12 weeks after the T-cell and/or vaccine infusion
  ORR defined as CR/PR/SD>6m (i.e., success = CR or PR or SD > 6m).

CONTACTS AND LOCATIONS:
Overall Officials: Rodabe N. Amaria, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saberian C, Amaria RN, Najjar AM, Radvanyi LG, Haymaker CL, Forget MA, Bassett RL, Faria SC, Glitza IC, Alvarez E, Parshottam S, Prieto V, Lizee G, Wong MK, McQuade JL, Diab A, Yee C, Tawbi HA, Patel S, Shpall EJ, Davies MA, Hwu P, Bernatchez C. Randomized phase II trial of lymphodepletion plus adoptive cell transfer of tumor-infiltrating lymphocytes, with or without dendritic cell vaccination, in patients with metastatic melanoma. J Immunother Cancer. 2021 May;9(5):e002449. doi: 10.1136/jitc-2021-002449. PMID 34021033
- [Derived] Joseph RW, Peddareddigari VR, Liu P, Miller PW, Overwijk WW, Bekele NB, Ross MI, Lee JE, Gershenwald JE, Lucci A, Prieto VG, McMannis JD, Papadopoulos N, Kim K, Homsi J, Bedikian A, Hwu WJ, Hwu P, Radvanyi LG. Impact of clinical and pathologic features on tumor-infiltrating lymphocyte expansion from surgically excised melanoma metastases for adoptive T-cell therapy. Clin Cancer Res. 2011 Jul 15;17(14):4882-91. doi: 10.1158/1078-0432.CCR-10-2769. Epub 2011 Jun 1. PMID 21632855
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org